CLINICAL TRIAL: NCT03646461
Title: A Multi-Institutional, Open-Label, Randomized, Phase II Trial Of Ibrutinib In Combination With EGFR Inhibition Or PD-1 Inhibition In Patients With Recurrent/Metastatic Head And Neck Squamous Cell Carcinoma
Brief Title: Trial of Ibrutinib Combined With Nivolumab or Cetuximab to Treat Recurrent/Metastatic HNSCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Principal Investigator, Kathryn Gold, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 161755
Record Dates: First submitted 2018-06-08; First posted 2018-08-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of the Head and Neck
Keywords: oropharyngeal
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — ibrutinib; Cetuximab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Open-label, multi-center, randomized, controlled, clinical trial. Enrollment will be stratified by HPV status and randomized in a 1:1 ratio to either ibrutinib + cetuximab or ibrutinib + nivolumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Ibrutinib + Cetuximab (Experimental): Ibrutinib 560mg PO daily (Imbruvica) PLUS Cetuximab 400mg/m2 x 1 then 250 mg/m2 weekly 28 day cycle
  Interventions: Drug: Ibrutinib 560mg PO daily (Imbruvica); Drug: Cetuximab
- Arm B: Ibrutinib + Nivolumab (Experimental): Ibrutinib 560mg PO daily (Imbruvica) PLUS Nivolumab 3mg/kg biweekly 28 day cycle
  Interventions: Drug: Ibrutinib 560mg PO daily (Imbruvica); Drug: Nivolumab

INTERVENTIONS:
Drug: Ibrutinib 560mg PO daily (Imbruvica) — BTK inhibitor combined with PD-1 inhibitor
  Other Names: Imbruvica
Drug: Cetuximab — Cetuximab 400mg/m2 x 1 then 250 mg/m2 weekly 28 day cycle
  Other Names: Erbitux
  Arms: Arm A: Ibrutinib + Cetuximab
Drug: Nivolumab — Nivolumab 3mg/kg biweekly 28 day cycle
  Other Names: opdivo
  Arms: Arm B: Ibrutinib + Nivolumab

SUMMARY:
This is an open-label, randomized, phase II trial to test the efficacy of Ibrutinib in combination with either Nivolumab or Cetuximab in the treatment of recurrent and/or metastatic head an neck squamous cell carcinoma

DETAILED DESCRIPTION:
Open-label, randomized, controlled, clinical trial. Enrollment will be stratified by HPV status and randomized in a 1:1 ratio to either ibrutinib + cetuximab or ibrutinib + nivolumab

The study will enroll patients who develop R/M HNSCC have not yet been treated with EGFR inhibitors in the recurrent/metastatic setting. All patients being considered for the study must be ≥ 18 years of age and will receive: i) ibrutinib + cetuximab or ii) ibrutinib + nivolumab.

To determine the clinical efficacy of ibrutinib in combination with cetuximab or nivolumab in patients with R/M HNSCC.

Ibrutinib will be supplied by Pharmacyclics as 140 mg hard gelatin capsules for oral (PO) administration.

Cetuximab will be supplied as a clear, colorless liquid formulated for intravenous administration.

Nivolumab will be supplied as a clear, colorless liquid formulated for intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

- To be enrolled in the study, each potential subject must satisfy all of the following inclusion criteria.

1. Histologically or cytologically proven squamous cell carcinoma of the head and neck not amenable to curative intent therapy. P16 or HPV status must be known on all patients with oropharyngeal primaries or unknown primaries.
2. Known p16 and/or HPV status by institutional standard.
3. Presence of measurable tumor lesions per RECIST criteria v1.1 by investigator review
4. Life expectancy greater than 12 weeks
5. Previously archived or newly obtained tumor specimens for correlative analysis
6. Adequate hematologic function independent of transfusion and growth factor support for at least 7 days prior to screening and randomization, with the exception of pegylated G-CSF (pegfilgrastim) and darbepoetin which require at least 14 days prior to screening and randomization defined as:

   * Absolute neutrophil count >750 cells/mm3 (0.75 x 109/L).
   * Platelet count >50,000 cells/mm3 (50 x 109/L).
   * Hemoglobin >8.0 g/dL.
7. Adequate hepatic and renal function defined as:

   * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN).
   * Estimated Creatinine Clearance ≥30 ml/min (Cockcroft-Gault)
   * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
8. PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN
9. Men and women ≥ 18 years of age.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
11. Female subjects who are of non-reproductive potential (ie, post-menopausal by history - no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry.
12. Male and female subjects who agree to use highly effective methods of birth control (eg, , implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence, or sterilized partner) and a barrier method (eg., condoms, vaginal ring, sponge, etc) during the period of therapy and for for 30 days after the last dose of study drug for females and 90 days for males.Ability and willingness to provide written informed consent

Exclusion Criteria:

- To be enrolled in the study, potential subjects must meet NONE of the following exclusion criteria:

1. Prior therapy with an EGFR inhibitor in the recurrent or metastatic setting
2. Nasopharyngeal carcinoma histology
3. Known, clinically active central nervous system metastases (stable metastases permitted)
4. Chemotherapy ≤ 28 days prior to first administration of study treatment and/or monoclonal antibody (including immunotherapy) ≤16 weeks prior to first administration of study treatment.
5. Prior exposure to BTK inhibitor, PD-1 inhibitor, or PD-L1 inhibitor
6. History of other malignancies, except:

   * Malignancy treated with curative intent and with no known active disease present for ≥3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ without evidence of disease.
7. Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc., or chronic administration [>14 days] of >10 mg/day of prednisone) within 28 days of the first dose of study drug.
8. Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
9. Recent infection requiring systemic treatment that was completed ≤14 days before the first dose of study drug.
10. Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE v4.0), Grade ≤1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
11. Known bleeding disorders (eg, von Willebrand's disease) or hemophilia.
12. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
13. Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
14. Any uncontrolled active systemic infection.
15. Any history of interstitial lung disease.
16. Active autoimmune disease or other contraindication to PD-1 inhibition.
17. Major surgery within 4 weeks of first dose of study drug.
18. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
19. Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
20. Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
21. Concomitant use of warfarin or other Vitamin K antagonists.
22. Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor
23. Currently active, clinically significant hepatic impairment Child-Pugh Class B or C according to the Child-Pugh Classification
24. Lactating or pregnant.
25. Unwilling or unable to participate in all required study evaluations and procedures.
26. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Efficacy of Combined Therapies using RECIST v1.1 | 3 yrs
  The primary endpoint is the clinical efficacy of each combinatorial treatment regimen as defined by the best overall response rate (proportion of patients with a partial or complete response in tumor burden) using RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival | 3 yrs
  Progression-free survival (PFS), defined as the interval from the date of first dose of ibrutinib to disease progression or death from any cause
Overall Survival | 3 yrs
  Overall survival (OS), defined as the date of first dose of ibrutinib to the date of death from any cause.
Duration of Response | 3 yrs
  Duration of response is measured from the time measurement criteria are met for complete response or partial response (whichever is recorded) until the first date that recurrent or progressive is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started)
Safety as assessed by the frequency of adverse events per CTCAE v4.0 | 3 yrs
  Overall frequency and severity of adverse events per CTCAE v4.0.

OTHER OUTCOMES:
Measurement of Biomarkers | 3 yrs
  Assessment of biomarkers in response to protocol based therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Gold, MD, Principal Investigator — University of California San Diego, Moores Cancer Center
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No